CLINICAL TRIAL: NCT01615757
Title: Comparison of Ara-c 12 gm/m2 vs 18 gm/m2 Per Cycle for 3 Cycles Each as Consolidation in AML ; An Open Label Randomized Non-inferiority Study
Brief Title: Safety and Efficacy Study of Ara-c at 18 gm/m2 Versus 12 gm/m2 for 3 Cycles Each in AML Consolidation
Acronym: Ara-c
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Prashant Mehta, Senior Resident , Department of Medical Oncology, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AML HIDAC, AIIMS
Record Dates: First submitted 2012-06-05; First posted 2012-06-11 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; Acute Myeloid Leukemia; Cytarabine dose; Ara-c dose; Consolidation
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm B, Ara-c - 12 gm/m2 (Experimental): Arm B will receive HIDAC at 12 gm/m2/cycle for 3 cycles , i.e. 2 gm/m2 BD , Day 1,3,5
  Interventions: Drug: Ara-c
- Arm A. Ara-c 18 gm/m2 (Active Comparator): Arm A will receive HIDAC at 18 gm/m2/cycle for 3 cycles , i.e. 3 gm/m2 BD , Day 1,3,5
  Interventions: Drug: Ara-c

INTERVENTIONS:
Drug: Ara-c — IV formulation, administered as a 2 hr infusion in 1 pint of normal saline, BD on D1,3,5 at 3 gm/m2 /dose
  Other Names: Cytosar, Cytarabine
  Arms: Arm A. Ara-c 18 gm/m2
Drug: Ara-c — IV formulation, administered as a 2 hr infusion in 1 pint of normal saline, BD on D1,3,5 at 2 gm/m2 /dose
  Other Names: Cytosar, Cytarabine
  Arms: Arm B, Ara-c - 12 gm/m2

SUMMARY:
The study will be conducted in the Department of Medical Oncology and Department of Haematology , AIIMS, Delhi. A total of 180 patients of Acute Myeloid Leukemia who are in complete remission after induction chemotherapy will be enrolled into the study and will be further randomized to the two study arms . ARM- A will receive Ara-c at 18 gm /m2 for 3 cycles and ARM -B will receive Ara-c at 12 gm/m2 for 3 cycles according to the study protocol. Aim of the study will be to compare the efficacy of the two doses in terms of the relapse free survival and overall survival as well as time to relapse and toxicity /treatment related morbidity.

DETAILED DESCRIPTION:
Objectives

* To compare the efficacy of two different doses of Cytarabine during consolidation therapy for newly diagnosed patients of Non APML - Acute Myeloid Leukemia who are in CR post induction
* To compare the toxicity of the two different Cytarabine doses

Primary end point

* Relapse free survival at 1 yr from randomization
* Relapse will be defined as >5 % leukemic blasts in the marrow aspirate or new extramedullary disease anytime after randomization

Secondary end points

* Overall survival
* Median time to relapse
* Toxicity- Haematological and Non -Haematological

Inclusion criteria

* Confirmation of Acute Myeloid Leukemia by morphologic, immunophenotypic analysis
* Suitable for HIDAC as consolidation
* AML with underlying MDS will be included

Exclusion criteria

* Previous AML chemotherapy [Hydroxyurea - not an exclusion.]
* CML-BC
* Concurrent active malignancy
* HIV infection, Uncontrolled Hepatitis B/C
* Patients being considered for upfront PBSCT (before completion of CONSOLIDATION)
* Serum Bilirubin > 2
* APML
* Delayed recovery of blood counts /persistent active infection > 45 days from start of induction
* Patients receiving reinduction with HIDAC
* Therapy related AML Methodology
* The period of enrollment will be from July 1, 2012 to September 30 ,2013
* Baseline information will be recorded in a preformulated proforma designed for analysis at a later date

Treatment

* Standard 3 + 7 INDUCTION with Daunomycin and Cytarabine with DNR at 60- 90 mg/m2 as per the PS and comorbidities/active infections at presentation
* Bone marrow examination - D+ 28 of induction or earlier if needed . Patients not in CR - reinduction regimen as per discretion of treating physician
* Patients in complete morphological remission ( after 1 or 2 inductions) : will receive consolidation with HIDAC and will be randomized into the two study arms after written Informed Consent: Arm A and B with 90 patients in each arm Arm A will receive HIDAC at 18 gm/m2/cycle for 3 cycles , i.e. 3 gm/m2 BD , Day 1,3,5 Arm B will receive HIDAC at 12 gm/m2/cycle for 3 cycles , i.e. 2 gm/m2 BD , Day 1,3,5

sample size

* Assuming a RFS of 60 % at 1 yr in each arm and keeping a non-inferiority margin of 20 % , Alpha at 5 % ,75 patients are required in each arm on the basis of statistical calculation.
* 15 patients added in each arm to account for losses
* Total required in each arm = 90
* ANC> 1000 , Platelet count > 1 lac required to start HIDAC
* Detailed information of the course of all the chemotherapy cycles will be recorded including-

  1. toxicity
  2. details of antimicrobials
  3. supportive care ( including transfusions)
  4. Use of growth factors
* Cytogenetic analysis using standard technique of chromosomal banding
* Molecular analysis for mutation of FLT3-ITD will be performed
* Risk stratification will be done as per guidelines
* Patients in both arms will be kept under close follow up and will be assessed with blood counts /PS , 2 monthly / or earlier as clinically indicated

Statistical Analysis

* Qualitative data will be analyzed using the Chi-square test
* Quantitative data will be compared by using t-test /Mann Whitney test
* Besides this survival analysis will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of Acute Myeloid Leukemia by morphologic, immunophenotypic analysis
* Suitable for HIDAC as consolidation
* AML with underlying MDS will be included

Exclusion Criteria:

* Previous AML chemotherapy [Hydroxyurea - not an exclusion.]
* CML-BC
* Concurrent active malignancy
* HIV infection, Uncontrolled Hepatitis B/C
* Patients being considered for upfront PBSCT (before completion of CONSOLIDATION)
* Serum Bilirubin > 2
* APML
* Delayed recovery of blood counts /persistent active infection > 45 days from start of induction
* Patients receiving reinduction with HIDAC
* Therapy related AML

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Relapse free survival at 1 yr of follow up | 1 year

SECONDARY OUTCOMES:
Toxicity- Haematological and Non -Haematological | at 1 yr
  The following variables will be compared in the two arms to -
  -Nadir blood counts,Ara c related fever ,Allergic or skin reactions,Alopecia,Diarrhea ,Stomatitis,Bleeding ,Febrile neutropenia,Infection(fungal /bacterial/viral),Liver related event,ocular toxicity,Neurologic event,Peripheral neuropathy,Cerebral/Cerebellar toxicity,Transfusions,Time to recovery of platelets,Time to recovery of neutrophils,Duration of Hospital stay,Emergency visits,Deaths,Use of growth factors

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Mehta, MD, Principal Investigator — AIIMS, Delhi, India; Vinod Raina, MD, Study Chair — AIIMS, Delhi
Locations (1):
- AIIMS, Delhi, National Capital Territory of Delhi, India